CLINICAL TRIAL: NCT03918265
Title: Tacrolimus Treatment for Refractory Autoimmune Cytopenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tacrolimus-2
Record Dates: First submitted 2019-04-16; First posted 2019-04-17 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-06

CONDITIONS: Autoimmune Hemolytic Anemia; Pure Red Cell Aplasia; Evans Syndrome
Keywords: Tacrolimus; Refractory autoimmune cytopenia; Prospective study
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Red-Cell Aplasia, Pure; Evans Syndrome | interventions — Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efficiency of tacrolimus on autoimmune cytopenia (Experimental): A prospective research of the tacrolimus efficiency on refractory autoimmune cytopenia patients. Dosage: 1mg bid and tacrolimus trough targets were 5-10 ng/ml throughout the study.
  Medication time should last at least 6 months.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — On refractory autoimmune cytopenia patients, tacrolimus was tried. Dosage: 1mg bid and tacrolimus trough targets were 5-10 ng/ml throughout the study
  Other Names: tacrolimus capsule

SUMMARY:
Autoimmune cytopenia, including autoimmune hemolytic anemia (AIHA), pure red cell aplasia (PRCA), Evans syndrome (ES), usually has good responses to steroids therapies as first line, but there is a considerable percentage of patients who relapse, become refractory or dependent on steroids to maintain an acceptable level of hemoglobin or platelets. The effects of the second line therapy are also not satisfactory and sometimes not available. The investigators aim to explore the efficacy and side-effect of tacrolimus for refractory autoimmune cytopenia.

DETAILED DESCRIPTION:
Tacrolimus binds FKBP12 with high affinity after entry into cytoplasm, suppresses calcineurin activity and prevents nuclear translocation of transcription factors such as NF-AT that are involved in IL-2 gene transcription. As a result, T-cell activation is inhibited with a subsequent reduction in the production of cytokines that include IL-2, TNF-α, IL-3, IL-4, IFN-γ, IL-6 and IL-10; B-cell activation, class-switching and immunoglobulin production are also attenuated. Reports on the use of tarcrolimus in the treatment of autoimmune cytopenia are anecdotal and describe therapy with a variety of drug dosages.

The purpose of this study is to evaluate the effect of tacrolimus on patients with refractory autoimmune cytopenia, the side-effects will be documented and plasma concentration of tacrolimus will be monitor.

ELIGIBILITY:
Inclusion Criteria:

* Refractory autoimmune cytopenia, including autoimmune hemolytic anemia, pure red cell aplasia, Evans syndrome.
* 18-80 years old.
* No response or intolerant to first and second line therapies.
* ECOG Performance Status of 0-2
* Written informed consent.

Exclusion Criteria:

* Other diseases which might cause hematological abnormalities.
* Response and well tolerate to first or second line therapy.
* Patients who are under 18-year-old or over 80-year-old.
* Pregnant or lactating.
* Patients unwilling to or unable to comply with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-04 (Actual); Primary Completion 2020-08-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | 6 months
  Hemoglobin level in g/L
Platelet count | 6 months
  Platelet count in /L

SECONDARY OUTCOMES:
Hemoglobin level | 2 years
  Hemoglobin level in g/L
Platelet count | 2 years
  Platelet count in /L

CONTACTS AND LOCATIONS:
Overall Officials: Bing Hang, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Feng X. Efficacy and safety of tacrolimus in systemic lupus erythematosus patients with refractory thrombocytopenia: a retrospective study. Lupus. 2018 Jan;27(1):60-65. doi: 10.1177/0961203317711011. Epub 2017 May 31. PMID 28566017
- [Background] Tabchi S, Hanna C, Kourie HR, Aftimos P, El Osta L, Ghosn M. Successful treatment of Evans syndrome with Tacrolimus. Invest New Drugs. 2015 Feb;33(1):254-6. doi: 10.1007/s10637-014-0155-9. Epub 2014 Sep 12. No abstract available. PMID 25209619